CLINICAL TRIAL: NCT01813877
Title: Randomized Metabolic Response Monitoring Trial in Patients With Suspected Recurrence of Glioblastoma F-DOPA PET/CT
Brief Title: Response Monitoring Trial in Patients With Suspected Recurrence of Glioblastoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: Kaiser Permanente (Other); The Methodist Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 12-000939; NCI-2013-01421 (Registry Identifier: CTRP); FDOPA12-000939 (Other: Jonsson Comprehensive Cancer Center)
Record Dates: First submitted 2013-03-07; First posted 2013-03-19 (Estimated); Last update posted 2020-07-27 (Actual); Status verified 2020-05

CONDITIONS: Glioma; Glioblastoma
MeSH Terms: conditions — Glioma; Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Diagnostics without PET (No Intervention)
- Diagnostics with PET (Experimental): All 18F-DOPA PET/CT studies will be interpreted qualitatively during a clinical readout session. Based on a previous study scans will be classified as positive if tumor regions defined on CT exhibited tracer uptake above the level of the contra-lateral caudate nucleus. Scans will be classified as negative if tumor 18F-FDOPA uptake is lower than that of the contra lateral caudate nucleus. Uptake at the level of the contra-lateral caudate will be considered equivocal for malignancy.
  Interventions: Radiation: FDOPA PET/CT

INTERVENTIONS:
Radiation: FDOPA PET/CT — Positron emission tomography (PET) is an established imaging technique that utilizes small amounts of radioactivity attached to very minimal amounts of substances (tracers) that are injected via a hand or arm vein. These substances can track certain features of cancers that can be visualized by using the PET/CT scanner, in this instance the amino acid 18F-DOPA.
  Arms: Diagnostics with PET

SUMMARY:
It was previously shown that 18F-DOPA PET imaging results in intended management changes in 41% of brain tumor patients. However, its impact on patient outcome defined as survival, costs, and/or quality of life has not been demonstrated. Regulatory agencies require randomized trials to determine the impact of PET on patient management and outcome. In this study we hypothesize that the addition of 18F-DOPA PET will improve patient outcome by more accurately identifying presence or absence of tumor recurrence than conventional imaging.

DETAILED DESCRIPTION:
Malignant gliomas are aggressive primary brain tumors that almost always lead to rapid patient deterioration and death. Timely diagnosis of recurrent disease as well as accurate monitoring of therapeutic responses is critically important in glioblastoma patients.

Despite introduction of new treatment approaches patient prognosis is poor with less than half of the patients being progression-free during the first 6 months after diagnosis of disease recurrence (6-month-progression-free survival rates of 46%).

The current diagnostic standard of care for diagnosing and monitoring brain tumors is contrast-enhanced, multi-planar magnetic resonance imaging (MRI). However, the ability of MRI for early detection of disease recurrence or progression is limited. Moreover, determination of treatment responses is difficult since benign tissue changes after radiation and/or chemotherapy can have the appearance of tumor recurrence or progression on MRI. Positron emission tomography (PET) is an established imaging technique that utilizes small amounts of radioactivity attached to very minimal amounts of substances (tracers) that are injected via a hand or arm vein. These substances can track certain features of cancers that can be visualized by using the PET/CT scanner. For instance, a number of different PET-tracers have been used to study brain tumor metabolism and to detect primary or recurrent tumors. These include tracers of glucose (18F-FDG) and amino acid metabolism (e.g. 18F-DOPA). Metabolic imaging of brain tumors with amino acid analogues has advantages over 18F-FDG. Since FDG assess glucose metabolism and the normal brain consumes a lot of glucose it can be difficult to detect tumors against high glucose use of normal brain tissue. 18FDOPA has been successfully used clinically for many years. The advantage of 18F-DOPA is that normal brain tissue consumes very little 18F-DOPA. Thus, tumors can be seen easily against a low background activity.

18F-DOPA PET imaging detects brain tumors with a very high accuracy and 18F-DOPA imaging affects the management of 40% of patients. However, its impact on patient outcome defined as survival, costs, and/or quality of life has not been demonstrated.

Randomized trials are needed to evaluate the impact of PET on patient management and outcome. We will determine this by randomizing patients with suspected recurrence of glioblastoma into those who are managed using conventional diagnostic imaging versus those who will receive conventional imaging plus 18F-DOPA PET. Randomization is like flipping a coin. Patients will have a 50% chance to undergo standard imaging or standard imaging combined with 18F-DOPA PET.

Approximately 25-40% of the patients with suspected tumor recurrence will have pseudo-progression on MRI (i.e. the images suggest that there is tumor recurrence when there is in fact no recurrence). These patients will have correctly negative 18F-DOPA PET scans. In these patient initiation of treatment can be postponed. In contrast, patients with positive 18F-DOPA PET scans will undergo some kind of treatment at the discretion of the treating physician (radiation therapy, chemotherapy or surgery). We will find out whether the management and treatment change that is based on 18FDOPA PET affects the survival of patients and affects the costs of caring for the patients.

ELIGIBILITY:
Inclusion Criteria:

* Suspected first recurrence of a glioblastoma tumor by clinical measures and/or MRI
* Age 18-99 years

Exclusion Criteria:

* Breast feeding/ Pregnancy
* Severe psychiatric illness
* Primary diagnosis of a glioblastoma

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2012-08-22 (Actual); Primary Completion 2020-01-14 (Actual); Study Completion 2020-01-14 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy compared to standard diagnostics without PET | 5 years
  Imaging findings will be validated by histopathology, clinical follow-up and/or repetitive imaging. If no histopathology within 3 months is available, clinical follow-up and imaging findings will be used for validation. If within 6 months of randomization no clinical progression nor progression on other imaging modalities is found, the patient will be rated as "no disease present at time of imaging".

SECONDARY OUTCOMES:
Impact of FDOPA PET on patient management | 7 years
  Overall and progression free survival will be assessed according to the standard of clinical care with a minimum follow-up time of two years after randomization. In this study protocol there are no pre-set follow-up algorithms, however in clinical routine a follow-up every three months is standard.

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Czernin, MD, Principal Investigator — Professor
Locations (1):
- UCLA, Los Angeles, California, United States

REFERENCES:
- See also: Ahmanson Imaging Division — http://www.pet.ucla.edu